CLINICAL TRIAL: NCT00040742
Title: A Phase II/III Randomized, Controlled Clinical Trial Of Ginger (Zingiber Officinale) For Nausea Caused By Chemotherapy For Cancer
Brief Title: Ginger in Treating Nausea in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC CCOP Research Base, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000069401; U10CA037420 (NIH); URCC U1902 (Other: University of Rochester CCOP Research Base); URCC-0114 (Other: NCI DCP)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Nausea; Vomiting
Keywords: nausea; vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Patients receive oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  Interventions: Other: placebo
- 0.5g ginger (Experimental): Patients receive oral low-dose ginger and oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  Interventions: Dietary Supplement: ginger; Other: placebo
- 1.0g ginger (Experimental): Patients receive oral intermediate-dose ginger and oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  Interventions: Dietary Supplement: ginger; Other: placebo
- 1.5g ginger (Experimental): Patients receive oral high-dose ginger twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  Interventions: Dietary Supplement: ginger

INTERVENTIONS:
Dietary Supplement: ginger — Given orally
  Arms: 0.5g ginger; 1.0g ginger; 1.5g ginger
Other: placebo — Given orally
  Arms: 0.5g ginger; 1.0g ginger; Placebo

SUMMARY:
RATIONALE: Ginger may help reduce or prevent nausea. It is not yet known if antiemetic drugs are more effective with or without ginger in treating nausea caused by chemotherapy.

PURPOSE: This randomized phase II/III trial is studying giving antiemetic drugs together with ginger to see how well they work compared to antiemetic drugs alone in treating nausea in patients who are receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of 1 course of ginger vs placebo when administered in regimens containing a 5-hydroxytryptamine type 3 (5-HT3) receptor antagonist antiemetic and dexamethasone (or the equivalent dose of IV methylprednisolone) in controlling chemotherapy-related nausea at course 2 of chemotherapy in patients with cancer.
* Compare the efficacy of 3 different doses of ginger in controlling chemotherapy-related nausea in these patients.
* Determine the adverse effects of ginger when given 3 days before chemotherapy administration in these patients.
* Determine the adverse effects of these antiemetic regimens during the 4 days after chemotherapy.
* Compare the chemotherapy-related anticipatory nausea in patients treated with these antiemetic regimens.
* Compare the quality of life during the 4 days after chemotherapy in patients treated with these antiemetic regimens.
* Compare the chemotherapy-related nausea at course 3 of chemotherapy in these patients after 2 courses of ginger vs placebo.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 4 treatment arms. Day 1 of each course is defined as the day of chemotherapy administration.

* Placebo: Patients receive oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
* 0.5g Ginger: Patients receive oral low-dose ginger and oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
* 1.0g Ginger: Patients receive oral intermediate-dose ginger and oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
* 1.5g Ginger: Patients receive oral high-dose ginger twice daily on days -3 to 3 of chemotherapy courses 2 and 3.

Patients in each arm also continue receiving their scheduled antiemetic regimen comprising a 5-hydroxytryptamine type-3 (5-HT3) receptor antagonist (ondansetron, granisetron, tropisetron, and dolasetron mesylate) and dexamethasone (DM) (or the equivalent dose of IV methylprednisolone (MePRDL)) on day 1 of courses 2 and 3.

Symptoms are assessed on day -3 to day 1 of courses 2 and 3 and on days 1-4 of courses 1-3.

Quality of life is assessed on day 4 of courses 1-3.

Nausea and vomiting are assessed 4 times daily on days 1-4 of courses 1-3.

PROJECTED ACCRUAL: A total of 706 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer and be scheduled to receive at least 3 courses of chemotherapy

  * Scheduled to receive chemotherapy with no planned interruption by radiotherapy or surgery
  * Chemotherapy courses must be separated by at least 2 weeks from day 1 to day 1 of next course
* Must have experienced nausea of any degree of severity after completion of the first study-related course of chemotherapy
* Received a prior 5-hydroxytryptamine type 3 (5-HT3) receptor antagonist antiemetic (ondansetron, granisetron, tropisetron, or dolasetron mesylate) with dexamethasone (DM) given at any dose and by any route (or equivalent dose of IV methylprednisolone (MePRDL)) on day 1 of course 1 of chemotherapy
* Scheduled to receive a 5-HT3 receptor antagonist antiemetic with DM (or equivalent dose of IV MePRDL) on day 1 of courses 2 and 3 of chemotherapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm^3 at second course of chemotherapy
* No prior bleeding or blood coagulation disorder (e.g., thrombocytopenia or platelet dysfunction)

Hepatic:

* No prior coagulation factor deficiency

Renal:

* Not specified

Cardiovascular:

* No prior vascular defect

Other:

* Able to understand English
* No concurrent or impending bowel obstruction

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent interferon therapy

Chemotherapy:

* See Disease Characteristics
* At least 6 months since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No concurrent warfarin or heparin for therapeutic anticoagulation
* Concurrent low-dose warfarin for maintenance of venous access allowed
* Concurrent rescue medications for control of symptoms caused by the cancer or its treatment allowed as clinically indicated

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 745 (Actual)
Dates: Start 2003-03; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L. Ryan, PhD, MPH, Study Chair — University of Rochester
Locations (19):
- United States (19):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhassett, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5g Ginger: Patients receive oral low-dose ginger and oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  ginger extract: Given orally
  placebo: Given orally
- 1.0g Ginger: Patients receive oral intermediate-dose ginger and oral placebo twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  ginger extract: Given orally
  placebo: Given orally
- 1.5g Ginger: Patients receive oral high-dose ginger twice daily on days -3 to 3 of chemotherapy courses 2 and 3.
  ginger extract: Given orally
Period: Overall Study
Arm/Group | Placebo | 0.5g Ginger | 1.0g Ginger | 1.5g Ginger
Started | 188 | 183 | 187 | 186 (One subject found to be ineligible after randomization. No baseline data collected.)
Completed | 149 | 134 | 141 | 152
Not Completed | 39 | 49 | 46 | 34
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Adverse Event | 15 | 16 | 21 | 9
Not completed — Withdrawal by Subject | 7 | 15 | 10 | 13
Not completed — Chemotoxicity | 4 | 3 | 5 | 2
Not completed — Incomplete Forms | 6 | 10 | 4 | 5
Not completed — Other medical | 7 | 5 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.5g Ginger | 1.0g Ginger | 1.5g Ginger | Total
Number analyzed (Participants) | 149 | 134 | 141 | 152 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10.62) | 54 (11.58) | 52 (10.69) | 52 (9.86) | 52.75 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 122 | 122 | 142 | 521
  Male | 14 | 12 | 19 | 10 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  White | 137 | 126 | 133 | 142 | 538
  Non-White | 11 | 8 | 7 | 10 | 36
  Unknown | 1 | 0 | 1 | 0 | 2
Education [Number; unit: participants]
  College Grad | 60 | 47 | 55 | 54 | 216
  H.S. Grad | 82 | 78 | 81 | 95 | 336
  Some/No HS | 6 | 9 | 5 | 3 | 23
  Unknown | 1 | 0 | 0 | 0 | 1
Previous surgery [Number; unit: participants]
  Yes | 131 | 115 | 126 | 129 | 501
  No | 18 | 19 | 15 | 23 | 75
Previous chemotherapy [Number; unit: participants]
  Yes | 81 | 75 | 85 | 82 | 323
  No | 68 | 57 | 56 | 70 | 251
  Unknown | 0 | 2 | 0 | 0 | 2
Previous radiation therapy [Number; unit: participants]
  Yes | 13 | 7 | 13 | 8 | 41
  No | 136 | 125 | 128 | 144 | 533
  Unknown | 0 | 2 | 0 | 0 | 2
Tumor site [Number; unit: participants]
  Alimentary | 14 | 11 | 10 | 8 | 43
  Breast | 107 | 100 | 103 | 117 | 427
  Genitourinary | 2 | 3 | 3 | 2 | 10
  Gynecologic | 11 | 6 | 9 | 5 | 31
  Hematologic | 3 | 4 | 9 | 8 | 24
  Lung | 10 | 7 | 6 | 10 | 33
  Other | 2 | 3 | 1 | 2 | 8
Marital status [Number; unit: participants]
  Married | 107 | 96 | 103 | 114 | 420
  Not Married | 42 | 38 | 38 | 38 | 156
Baseline average nausea, Day1 [Mean (Standard Deviation); unit: units on a scale] — Average nausea evaluated using a 7-point semantic rating scale anchored by "1" = " Not at all nauseated" and by "7" = "Extremely nauseated."
  units on a scale | 2.2 (1.6) | 2.6 (1.9) | 2.5 (1.8) | 2.4 (1.7) | 2.4 (1.8)
Baseline nausea at its worst [Mean (Standard Deviation); unit: units on a scale] — Maximum nausea evaluated using a 7-point semantic rating scale anchored by "1" = " Not at all nauseated" and by "7" = "Extremely nauseated."
  units on a scale | 2.5 (1.7) | 2.9 (2.1) | 2.8 (2.0) | 2.7 (2.0) | 2.7 (2.0)
Quality of life(FACT-G) [Mean (Standard Deviation); unit: units on a scale] — Quality of life is evaluated using the Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item compilation of questions divided into 4 primary domains: Physical Well-Being (PWB)[range 0 - 28], Social Well-Being (SWB)[range 0 - 28], Emotional Well-Being (EWB) [range 0 - 24], and Functional Well-Being (FWB) [range 0 - 28]. Total FACT-G score is a sum of the 4 primary domains [range 0 - 108]. The higher the score, the better.
  units on a scale | 72 (15.9) | 72 (15.0) | 71 (15.4) | 72 (16.0) | 72 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Peak Acute Nausea
Description: Nausea evaluated on a 7-point semantic rating scale anchored by "1" = "Not at all nauseated" and by "7" = "Extremely nauseated." Acute nausea calculated as the maximum of the Day 1 Evening and Night nausea ratings.
  Change from post-intervention (cycle 2 of chemotherapy) - baseline (cycle 1 of chemotherapy) of peak acute nausea used as the outcome measure.
  Negative values for this outcome are favorable.
Time Frame: 3-4 days on study drug
Population: Eligible patients 18 years of age or older, able to understand English, diagnosed with cancer, may have received more than one chemotherapy cycle and scheduled for at least three additional cycles; randomization stratified by CCOP site. A computer-generated random numbers table assigned patients to one of four treatment arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 0.5g Ginger | 1.0g Ginger | 1.5g Ginger
Number analyzed (Participants) | 149 | 134 | 141 | 152
units on a scale | 0.03 (1.85) | -0.56 (1.83) | -0.44 (1.79) | -0.15 (1.82)
Statistical Analysis 1: Comparison: Placebo vs 0.5g Ginger; H0: Mean difference between 0.5g and placebo of change from baseline of Peak Acute Nausea = 0. Ha: Mean difference between 0.5g and placebo of change from baseline of Peak Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = .017, Mixed Models Analysis — The p-value was adjusted using theTukey-Kramer method; Mixed model analyses and Type 3 tests of fixed effects using the Kenward-Roger degrees of freedom procedure were used; Mean Difference (Final Values) = -0.566, Standard Error of Mean 0.145 — The estimation parameter (mean difference) is the difference in mean change from baseline (post-intervention - baseline) between groups (0.5 gm ginger - placebo). Negative values are favorable for the ginger group
Statistical Analysis 2: Comparison: Placebo vs 1.0g Ginger; H0: Mean difference between 1.0g and placebo of change from baseline of Peak Acute Nausea = 0. Ha: Mean difference between 1.0g and placebo of change from baseline of Peak Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — The p-value was adjusted using theTukey-Kramer method; Mixed model analyses and Type 3 tests of fixed effects using the Kenward-Roger degrees of freedom procedure were used; Mean Difference (Final Values) = -0.506, Standard Error of Mean 0.141 — The estimation parameter (mean difference) is the difference in mean change from baseline (post-intervention - baseline) between groups (1 gm ginger - placebo). Negative values are favorable for the ginger group
Statistical Analysis 3: Comparison: Placebo vs 1.5g Ginger; H0: Mean difference between 1.5g and placebo of change from baseline of Peak Acute Nausea = 0. Ha: Mean difference between 1.5g and placebo of change from baseline of Peak Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.431, Mixed Models Analysis — The p-value was adjusted using theTukey-Kramer method; Mixed model analyses and Type 3 tests of fixed effects using the Kenward-Roger degrees of freedom procedure were used; Mean Difference (Final Values) = -0.269, Standard Error of Mean 0.137 — The estimation parameter (mean difference) is the difference in mean change from baseline (post-intervention - baseline) between groups (1.5 gm ginger - placebo). Negative values are favorable for the ginger group
Statistical Analysis 4: Comparison: Placebo vs 0.5g Ginger vs 1.0g Ginger vs 1.5g Ginger; Placebo vs. Any Ginger. H0: Mean difference between [(0.5g +1.0g +1.5g) / 3] and placebo of change from baseline of Peak Acute Nausea = 0. Ha: Mean difference between [(0.5g +1.0g +1.5g) / 3] and placebo of change from baseline of Peak Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Parameter estimated using a contrast; Mean Difference (Final Values) = -0.470, Standard Error of Mean 0.160 — The estimation parameter (mean difference) is the difference in mean change from baseline (post-intervention - baseline) between groups (any ginger - placebo). Negative values are favorable for the ginger group

2. Secondary Outcome: Average Nausea Severity
Description: Nausea evaluated on a 7-point semantic rating scale anchored by "1" = "Not at all nauseated" and by "7" = "Extremely nauseated." Acute nausea calculated as the average of the Day 1 Evening and Night nausea ratings.
  Change from post-intervention (cycle 2 of chemotherapy) - baseline (cycle 1 of chemotherapy) of average acute nausea used as the outcome measure.
  Negative values for this outcome are favorable.
Time Frame: 3-4 days on study drug
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.5g Ginger | 1.0g Ginger | 1.5g Ginger
Number analyzed (Participants) | 149 | 134 | 141 | 152
units on a scale | 0.03 (1.58) | -0.44 (1.67) | -0.34 (1.64) | -0.05 (1.68)
Statistical Analysis 1: Comparison: Placebo vs 0.5g Ginger; H0: Mean difference between 0.5g and placebo of change from baseline of Average Acute Nausea = 0. Ha: Mean difference between 0.5g and placebo of change from baseline of Average Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.046, Mixed Models Analysis — The p-value was adjusted using theTukey-Kramer method; Mixed model analyses and Type 3 tests of fixed effects using the Kenward-Roger degrees of freedom procedure were used; Mean Difference (Final Values) = -0.441, Standard Error of Mean 0.127 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 1.0g Ginger; H0: Mean difference between 1.0g and placebo of change from baseline of Average Acute Nausea = 0. Ha: Mean difference between 1.0g and placebo of change from baseline of Average Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.076, Mixed Models Analysis — The p-value was adjusted using theTukey-Kramer method; Mixed model analyses and Type 3 tests of fixed effects using the Kenward-Roger degrees of freedom procedure were used; Mean Difference (Final Values) = -0.402, Standard Error of Mean 0.124 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 1.5g Ginger; H0: Mean difference between 1.5g and placebo of change from baseline of Average Acute Nausea = 0. Ha: Mean difference between 1.5g and placebo of change from baseline of Average Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.738, Mixed Models Analysis — The p-value was adjusted using theTukey-Kramer method; Mixed model analyses and Type 3 tests of fixed effects using the Kenward-Roger degrees of freedom procedure were used; Mean Difference (Final Values) = -0.158, Standard Error of Mean 0.120 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 0.5g Ginger vs 1.0g Ginger vs 1.5g Ginger; Placebo vs Any Ginger. H0: Mean difference between [(0.5g +1.0g +1.5g) / 3] and placebo of change from baseline of Average Acute Nausea = 0. Ha: Mean difference between [(0.5g +1.0g +1.5g) / 3] and placebo of change from baseline of Average Acute Nausea > 0. (Two-sided); Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; Contrasts used for estimation; Mean Difference (Final Values) = -0.350, Standard Error of Mean 0.140 — [estimate comment as in outcome 1, analysis 4]

ADVERSE EVENTS:
Arm/Group | Placebo | 0.5g Ginger | 1.0g Ginger | 1.5g Ginger
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/183 | 1/187 | 0/187
Other Adverse Events (participants affected / at risk) | 5/188 | 7/183 | 3/187 | 8/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=188) | 0.5g Ginger (N=183) | 1.0g Ginger (N=187) | 1.5g Ginger (N=187)
Death (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=188) | 0.5g Ginger (N=183) | 1.0g Ginger (N=187) | 1.5g Ginger (N=187)
Gastrointestinal symptoms (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bruising/flushing, rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Blood disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebral disorders (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weakness, dizziness, fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Two main weaknesses of the study, which should be controlled for in future studies, were not controlling for chemotherapy regimens (i.e., high versus low emetogenic regimens) or the severity level of nausea before enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No